CLINICAL TRIAL: NCT06044558
Title: Effect of Azole/Echinocandin Use on Tacrolimus Pharmacokinetics in Kidney Transplant Recipients
Brief Title: Effect of Azole/Echinocandin Use on Tacrolimus Pharmacokinetics
Status: Completed | Type: Observational
Sponsor: LI YAN (Other)
Responsible Party: Sponsor-Investigator, LI YAN, director, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: QFS-LY-2023-TAC-001
Record Dates: First submitted 2023-08-28; First posted 2023-09-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Kidney Transplant Patients
Keywords: tacrolimus; voriconazole; C0/D; CYP3A5; drug-drug interactions; caspofungin; kidney transplant
MeSH Terms: interventions — Voriconazole; Tacrolimus; Methylprednisolone Hemisuccinate; Mycophenolic Acid; Caspofungin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Combined with voriconazole group: Methylprednisolone sodium succinate was administered intravenously the day after transplantation at an initial dose of 500 mg/day, with the dose being tapered evenly to 40 mg/day during the first week. During the second week, methylprednisolone tablets were administered continuously at a dose of 40 mg/day, after which the dose was tapered to 16 mg/day as a maintenance dose. Immunosuppression was maintained with oral mycophenolate sodium 720 mg twice daily. For renal transplant patients, the initial oral tacrolimus dose should be 0.15 - 0.30 mg/kg per day divided into morning and evening doses. The starting dose of voriconazole should be 400 mg twice a day, which should be changed to 200 mg twice a day from the next day as a maintenance dose.
  Interventions: Drug: Combined with voriconazole
- Combined with caspofungin group: Methylprednisolone sodium succinate was administered intravenously the day after transplantation at an initial dose of 500 mg/day, with the dose being tapered evenly to 40 mg/day during the first week. During the second week, methylprednisolone tablets were administered continuously at a dose of 40 mg/day, after which the dose was tapered to 16 mg/day as a maintenance dose. Immunosuppression was maintained with oral mycophenolate sodium 720 mg twice daily. For renal transplant patients, the initial oral tacrolimus dose should be 0.15 - 0.30 mg/kg per day divided into morning and evening doses. The dosage of caspofungin was 70 mg intravenous injection once on the first day after surgery and 50 mg intravenous injection once a day starting from the second day.
  Interventions: Drug: Combined with caspofungin
- Tacrolimus-alone treatment group: Methylprednisolone sodium succinate was administered intravenously the day after transplantation at an initial dose of 500 mg/day, with the dose being tapered evenly to 40 mg/day during the first week. During the second week, methylprednisolone tablets were administered continuously at a dose of 40 mg/day, after which the dose was tapered to 16 mg/day as a maintenance dose. Immunosuppression was maintained with oral mycophenolate sodium 720 mg twice daily. For renal transplant patients, the initial oral tacrolimus dose should be 0.15 - 0.30 mg/kg per day divided into morning and evening doses.
  Interventions: Drug: Tacrolimus-alone treatment

INTERVENTIONS:
Drug: Combined with voriconazole — Renal transplant patients taking tacrolimus-based triple immunotherapy and voriconazole drug combination.
  Other Names: tacrolimus; methylprednisolone sodium succinate; mycophenolate sodium
  Groups: Combined with voriconazole group
Drug: Combined with caspofungin — Renal transplant patients taking a combination of tacrolimus-based triple immunotherapy and caspofungin drugs.
  Other Names: tacrolimus; methylprednisolone sodium succinate; mycophenolate sodium
  Groups: Combined with caspofungin group
Drug: Tacrolimus-alone treatment — Renal transplant patients treated with tacrolimus-based triple immunotherapy alone
  Other Names: methylprednisolone sodium succinate; mycophenolate sodium
  Groups: Tacrolimus-alone treatment group

SUMMARY:
The purpose of this observational study is to analyze the extent and characteristics of drug interactions (focusing on azole antifungals and echinocandins) and genetic polymorphisms on tacrolimus blood concentrations in renal transplant recipients in order to provide a reference for the appropriate adjustment of tacrolimus dosing regimen to reduce the incidence of adverse drug reactions and rejection, and to improve the survival of transplanted kidneys.

DETAILED DESCRIPTION:
In this study, investigators investigated the effects of CYP3A5 and CYP2C19 gene polymorphisms on the trough concentration of tacrolimus after renal transplantation in recipients who were on a tacrolimus-based immunosuppressive regimen (tacrolimus + mescaline + glucocorticosteroid) after their first renal transplantation; investigators investigated the effects of antifungal drugs on the trough concentration of tacrolimus, and investigators also analyzed the effects of genetic factors on the drug-drug interactions between antifungal drugs and tacrolimus, with the aim of providing a basis of reference for the rational use of tacrolimus and antifungal drugs in the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with first kidney transplantation and intact CYP3A5 genotype;
2. Renal transplant recipients taking a tacrolimus-based triple immunosuppressive regimen (tacrolimus + sodium mescaline enteric-coated tablets + glucocorticoids) postoperatively;
3. Age ≥ 18 years.

Exclusion Criteria:

1. Missing and incomplete clinical information and postoperative follow-up data;
2. Multi-organ combined transplantation and secondary transplantation;
3. Postoperative simultaneous joint application of other drugs that affect the blood concentration of tacrolimus or voriconazole or caspofungin (e.g. pentoxifylline capsules, rifampicin, etc.);
4. Severe impairment of liver function or severe gastrointestinal diseases, gastrointestinal resection surgery, malabsorption syndrome;
5. Pregnant and lactating women;
6. Recipients with significant rejection of the transplanted organ or death due to other reasons within 1~2 months after surgery;
7. Poor compliance and accuracy of results (e.g., irregular blood collection times).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included patients who underwent renal transplantation at our hospital between 01.01.2015 and 04.01.2023 and were divided into the co-voriconazole group, co-carbophenazole group and tacrolimus alone group according to co-administration.
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
The C0/D values of tacrolimus | 2015.01.01-2023.04.01
  Body weight is in kilograms, D values are in mg/d, and the combination of body weight and D is the body weight-corrected D value in mg/kg/d, with a range of 0.15-0.30 mg/kg/d. The C0 for tacrolimus is in ng/ml, with a range of 5-15 ng/ml, and the combination of the C0 and body weight-corrected D values is the C0/D value, reported as (ng/ml)/(mg /kg/d) is reported.

SECONDARY OUTCOMES:
The D values of tacrolimus | 2015.01.01-2023.04.01
  Body weight was expressed in kilograms, D values were expressed in mg/d, and body weight and D were combined to give body weight-corrected D values in mg/kg/d, ranging from 0.15 to 0.30 mg/kg/d.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT06044558/Prot_SAP_002.pdf
  • Informed Consent Form (2023-02-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT06044558/ICF_003.pdf